CLINICAL TRIAL: NCT00159172
Title: Phase 1 Study of Motor Cortex Stimulation in the Treatment of Advanced Parkinson Disease
Brief Title: Safety and Efficacy of Motor Cortex Stimulation in the Treatment of Advanced Parkinson Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: Parkostim
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-03-06 (Estimated); Status verified 2005-09

CONDITIONS: Parkinson Disease
Keywords: Advanced parkinson disease; Stimulation; Motor Cortex; Parkinson disease C10.574.812; Electric Stimulation Therapy E02.831.580.438; Neuronavigation E05.873.249
MeSH Terms: conditions — Parkinson Disease

INTERVENTIONS:
Device: Motor cortex stimulation

SUMMARY:
The purpose of this study is to determine whether motor cortex stimulation, a mildly invasive surgical procedure, is safe and effective in advanced stage Parkinsonian patients who display side effects with dopaminergic treatment.

DETAILED DESCRIPTION:
Advanced stage of Parkinson disease (PD) is a difficult condition to treat, especially after several years of dopaminergic drugs. Recent development of neurosurgical techniques using deep brain stimulation leads has shown good behavioral results in these advanced PD patients. However, the placement of a stimulation lead in the subthalamic nucleus is a complex, invasive, and long surgical procedure. Such intervention requires a sophisticated technical environment, including a stereotactic magnetic resonance imaging (MRI) exam, associated with per-operative electrophysiological exploration of deep brain structures. This surgical treatment can therefore be indicated only for a few selected patients, and cannot be offered to a large proportion of patients among the potential candidates (estimation of 5000 patients in France). Thus, there is a need to develop therapeutic alternatives that would be technically and practically more convenient, less invasive, and that could be offered to a larger number of patients. Several clinical studies, including one led by our group, have already demonstrated that transcranial magnetic cortical stimulation could improve bradykinesia and shorten motor reaction time in patients with Parkinson disease. The clinical benefit was however moderate, and transient, probably because the stimulating sessions were too short in duration.

A prolonged effect could be obtained with continuous cortical stimulation. Such cortical stimulation has already been developed with good clinical tolerance in our hospital since 1991 for chronic neuropathic pain syndromes. In a non-human primate model of late stage Parkinson disease, we have recently demonstrated that prolonged primary motor cortex stimulation significantly improved both akinesia and bradykinesia.

The primary objective of this pilot study will be to evaluate the tolerance and efficacy of chronic stimulation of the primary motor cortex in 10 patients suffering from advanced stage Parkinson disease, despite the optimisation of dopaminergic treatment. The expected benefit for the patient will be gait improvement, increased movement velocities, and finally a better quality of life associated with reduction in dopaminergic medication and low per-operative morbidity risk.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Idiopathic Parkinson disease, for at least 5 years of evolution
* Asymmetric akinetic-rigid form, with symptoms predominant in the right side of the body (stimulator will be implanted on the left side).
* Functional impairment score in off stage (no drug treatment) of 3-4 according to the Hoehn and Yahr scale
* UPDRS III score > 40 in off-drug stage.
* UPDRS III score with L-dopa treatment improved by at least 50% compared to UPDRS III score in off-drug stage

Exclusion Criteria:

* Age superior to 70 years
* Adult patients under guardianship
* Previous neurosurgical operation(s)
* Previous partial or generalised seizures
* Mini Mental Status (MMS) score  24 or Mattis score < 130 or Montgomery-Asberg Depression Rating Scale (MADRS) depression score > 20.
* Presence of signal abnormalities on T1- and T2- MRI sequences
* Abnormalities in general exam or biological constants (hemogram, ionogram, hepatic or kidney dysfunction) with a higher surgical risk

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2005-09; Study Completion 2008-05

PRIMARY OUTCOMES:
Safety of the treatment and Unified Parkinson Disease Rating Scale (UPDRS) III 1 month following constant stimulation with and without motor cortex stimulation when the patient has no anti-parkinsonian drug for 12 hours

SECONDARY OUTCOMES:
Quality of life: Parkinson's Disease Questionnaire 39 (PDQ39) scores
Anti-parkinsonian drug doses (equivalent L-dopa)
Results of motor activation study in positron emission tomography (PET) scan
Results of the different neuropsychological tests
Video movement analysis

CONTACTS AND LOCATIONS:
Overall Officials: Stephane Palfi, MD, PhD, Principal Investigator — Paris 12 University- APHP
Locations (1):
- Neurosurgical Department Henri Mondor Hospital, Créteil, France

REFERENCES:
- [Background] Drouot X, Oshino S, Jarraya B, Besret L, Kishima H, Remy P, Dauguet J, Lefaucheur JP, Dolle F, Conde F, Bottlaender M, Peschanski M, Keravel Y, Hantraye P, Palfi S. Functional recovery in a primate model of Parkinson's disease following motor cortex stimulation. Neuron. 2004 Dec 2;44(5):769-78. doi: 10.1016/j.neuron.2004.11.023. PMID 15572109